CLINICAL TRIAL: NCT02602691
Title: Cost-utility Analysis of the AlloMap® Test for the Monitoring of Patients After Heart Transplantation
Brief Title: Cost-utility Analysis of the AlloMap® Test
Acronym: CUPIDON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL14_0455; IDRCB (Other: 2015-A00808-41)
Record Dates: First submitted 2015-11-09; First posted 2015-11-11 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Heart Transplantation
Keywords: Heart transplantation; AlloMap® gene expression profiling test; Medico-economic study

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Endomyocardial biopsy (Active Comparator): Systematic endomyocardial biopsies performed according to a planned monitoring schedule in usual care for patients with a heart transplantation.
  Interventions: Procedure: Endomyocardial biopsies
- AlloMap® test (Experimental): Noninvasive gene expression profiling blood test (AlloMap®) performed instead of endomyocardial biopsies when planned in the monitoring schedule for patients with a heart transplantation.
  Interventions: Other: AlloMap®

INTERVENTIONS:
Other: AlloMap®
  Arms: AlloMap® test
Procedure: Endomyocardial biopsies
  Arms: Endomyocardial biopsy

SUMMARY:
Transplant rejection is one of the most important complications of heart transplantation and requires a specific monitoring, including regular and invasive endomyocardial biopsies.

The average hospital cost of a biopsy has been estimated at 3 297 dollars in United States. In France, the reimbursement rates by the Health Insurance for the corresponding stays vary from 682 to 25 865 euros, according to the finding of a rejection and its severity.

AlloMap® is a non-invasive blood test that can identify patients with low probability of moderate to severe acute cell transplant rejection. The non-inferiority of the use of the AlloMap® test has been demonstrated in comparison of the usual care in terms of diagnosis of acute cellular rejection in a randomized study conducted in the United States. Following this study, the ISHLT (International Society of Heart and Lung Transplantation) made recommendations advocating its use for these patients between 6 months and 5 years after heart transplantation. This new test could be an alternative to systematic biopsies usually performed to patients whose allograft function is stable, but it is very expensive since the analysis of a blood sample cost 2 000 euros pre-tax in France. This cost has to be compared with the current patient care. By replacing biopsies performed systematically, the test should reduce the costs of full and day hospitalizations for the realization of biopsies but also the costs associated with their possible complications. In addition, it can be expected that its use provides a benefit to the patient in terms of quality of life. Indeed, the achievement of a biopsy may cause significant stress and anxiety for the patient, due to discomfort, pain and potential complications that may be severe.

To this day, no medico-economic assessment has been conducted to prove the interest of the use of AlloMap® compared to systematic realization of endomyocardial biopsies. The purpose of the CUPIDON study is to assess the effectiveness of the use of the AlloMap® test for monitoring heart transplant patients in the context of usual care and in accordance with international recommendations. AlloMap® will be used and compared to the current surveillance strategy by endomyocardial biopsies from 6 months to 36 months after heart transplantation. The investigators hypothesize that the use of this test for the diagnosis of acute cellular transplant rejection would avoid the costs of a large number of biopsies, while increasing the quality of life of patients related to their health.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Heart transplantation since 5 months (+/- 3 weeks)
* Stable allograft function :

  * Left ventricular ejection fraction ≥ 50% measured by echocardiography
  * No sign of the presence of humoral rejection or DSA (donor-specific antibodies)
  * Absence of biopsy-proven or treated acute cellular rejection in the previous 3 months
* Signed consent to participate in the study
* Patient affiliated to a social security scheme or similar

Exclusion Criteria:

* All symptoms or clinical signs of graft failure
* Treatment of a transplant rejection with ISHLT grade 2R or higher (proven by biopsy) during the previous 3 months
* Change of immunosuppressive molecule in the previous 30 days
* Treatment with hematopoietic growth factors in progress or during the previous 30 days
* Corticosteroid dose > 20 mg / day prednisone equivalent at the time of inclusion
* Transfusion during the previous 30 days
* End-stage renal failure requiring renal replacement therapy (hemodialysis or peritoneal dialysis)
* Pregnant woman at the time of inclusion
* Major patient protected by law

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2022-10-28 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
Incremental cost per quality-adjusted life-years (QALY) between systematic biopsies and use of the gene expression profiling blood test AlloMap® in monitoring of heart transplant patients for rejection | 36 months after heart transplantation
  QALY will be measured using the EQ-5D quality of life questionnaire. The cost analysis will be conducted from the viewpoints of the French Health Insurance and the hospital, considering only hospital direct costs. All resource consumption, outside the AlloMap® test, will be commonly valued by standard costs.

SECONDARY OUTCOMES:
Budget Impact analysis: estimation of the cost difference of the care of heart transplant patients before and after the introduction of the AlloMap® test | 36 months after heart transplantation
  Estimation of the cost difference of the care of heart transplant patients from the viewpoint of the French Health Insurance between two situations:
  * The current situation before the introduction of the innovative strategy: to estimate the overall cost in monitoring of heart transplant patients in France.
  * A hypothetical situation after the introduction of the innovative strategy: the impact of the introduction of the innovative strategy in the care of heart transplant patients must be simulated and the cost for this new situation must be estimated.
Quality of life | At inclusion visit (5 months after heart transplantation)
  Quality of life coefficient will be estimated with the EQ-5D questionnaire
Quality of life | At 12 months after heart transplantation
  Quality of life coefficient will be estimated with the EQ-5D questionnaire
Quality of life | At 18 months after heart transplantation
  Quality of life coefficient will be estimated with the EQ-5D questionnaire
Quality of life | At 24 months after heart transplantation
  Quality of life coefficient will be estimated with the EQ-5D questionnaire
Quality of life | At 30 months after heart transplantation
  Quality of life coefficient will be estimated with the EQ-5D questionnaire
Quality of life | At 36 months after heart transplantation
  Quality of life coefficient will be estimated with the EQ-5D questionnaire
Number of endomyocardial biopsies between the sixth and the thirty-sixth months after heart transplantation | 30 months
Number and types of complications secondary to endomyocardial biopsies between the sixth and the thirty-sixth months after heart transplantation | 30 months
Number of treated cell transplant rejection between the sixth and the thirty-sixth months after heart transplantation | 30 months
  Global number and number per ISHLT grade
Number of treated humoral transplant rejection between the sixth and the thirty-sixth months after heart transplantation | 30 months
Number of transplant rejection with hemodynamic consequences between the sixth and the thirty-sixth months after heart transplantation | 30 months
Number of transplant rejection proven by endomycardial biopsy between the sixth and the thirty-sixth months after heart transplantation | 30 months
Global survival | 36 months after heart transplantation
Survival without transplant rejection | 36 months after heart transplantation
Survival without graft dysfunction | 36 months after heart transplantation
  Dysfunction will be defined with ejection fraction ≤30% on echocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Laurent SEBBAG, MD, Principal Investigator — Hospices Civils de Lyon
Locations (13):
- France (13):
  - CHU, Hôpital du Haut Lévèque, Bordeaux
  - CHU, Hôpital Michallon, La Tronche
  - CHRU de Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - CHU, Hôpital La Timone, Marseille
  - CHU A. de Villeneuve, Montpellier
  - CHU, Hôpital Nord Laennec, Nantes
  - AP-HP, Hôpital Bichat, Paris
  - AP-HP, Hôpital La Pitié Salpêtrière, Paris
  - CHU de Rennes, Rennes
  - CHU, Hôpital Charles Nicolle, Rouen
  - CHRU de Strasbourg, Strasbourg
  - CHU, Hôpital Rangueil, Toulouse